CLINICAL TRIAL: NCT00070083
Title: A Phase I Study Of G3139 Antisense Oligonucleotide (Oblimersen) In Combination With CHOP And Rituximab In Untreated Advanced Stage Diffuse Large B Cell Lymphoma
Brief Title: Oblimersen, Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Treating Patients With Stage II, Stage III, or Stage IV Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000329985; BCCA-NCI-5818; NCI-5818
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2005-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — oblimersen; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

INTERVENTIONS:
Biological: oblimersen sodium
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, use different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of a chemotherapy drug by making cancer cells more sensitive to the drug. Combining oblimersen with rituximab and combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of oblimersen when given together with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone in treating patients with stage II, stage III, or stage IV large B-cell lymphoma

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and safety of oblimersen administered in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone, in terms of short-term and long-term toxicity, in patients with previously untreated stage III or IV or extensive or bulky stage II diffuse large B-cell lymphoma.
* Determine the maximum tolerated dose of oblimersen administered with this regimen in these patients.

Secondary

* Determine the remission rate and failure-free, progression-free, and overall survival of patients treated with this regimen.

OUTLINE: This is a nonrandomized, non-blinded, multicenter, dose-escalation study of oblimersen.

Patients receive CHOP-R* therapy comprising cyclophosphamide IV over 15-45 minutes, doxorubicin IV over 5-10 minutes, vincristine IV, and rituximab IV over 30-90 minutes on day 1 and oral prednisone on days 1-5. Patients also receive oblimersen IV continuously on days -4 to 3. Treatment repeats every 21 days for 6-8 courses in the absence of disease progression or unacceptable toxicity. Patients who discontinue treatment due to unacceptable toxicity to oblimersen may continue to receive standard therapy comprising CHOP-R.

NOTE: *Patients treated at the British Columbia Cancer Agency receive cyclophosphamide, doxorubicin, vincristine, and rituximab on days 1 and 2 and prednisone as above.

Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 10 patients are treated at that dose level.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-28 patients will be accrued for this study within 5-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* CD20+ diffuse large B-cell lymphoma, including any of the following stages:

  * Extensive stage II (not radio-encompassable within a single involved field or not a candidate for brief chemotherapy and radiotherapy)
  * Bulky stage II (any single mass greater than 10 cm)
  * Stage III
  * Stage IV NOTE: *Confirmed by tissue biopsy
* Previously untreated disease
* Measurable disease

  * At least 2 cm by imaging studies
* Circulating lymphoma cells no greater than 5,000/mm^3
* No history of other lymphoproliferative disorder
* No history of indolent lymphoma
* No T-cell lymphoma
* No CNS involvement
* No post-transplantation lymphoproliferative disorder

PATIENT CHARACTERISTICS:

Age

* 19 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3 (unless due to bone marrow involvement with lymphoma)
* Platelet count at least 100,000/mm^3 (unless due to splenomegaly or bone marrow involvement with lymphoma)

Hepatic

* Bilirubin no greater than 3 mg/dL (unless due to lymphoma)
* No known hepatitis B virus

Renal

* Creatinine no greater than 2 mg/dL (unless due to lymphoma)

Cardiovascular

* No cardiac contraindication to doxorubicin therapy (e.g., abnormal contractility on echocardiography)
* History of cardiac disease allowed provided ejection fraction is normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate venous access
* HIV negative
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer, localized basal cell or squamous cell skin cancer, or curatively treated carcinoma in situ of the cervix
* No neurological contraindication to vincristine (e.g., peripheral neuropathy)
* No active systemic infection
* No medical condition that would compromise study treatment, add toxicity, or impair assessment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

  * Prior radiotherapy for localized basal cell or squamous cell skin cancer used with curative intent allowed

Surgery

* Not specified

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Klasa, MD, Study Chair — British Columbia Cancer Agency
Locations (4):
- Stanford Cancer Center at Stanford University Medical Center, Stanford, California, United States
- Canada (3):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia